CLINICAL TRIAL: NCT07062458
Title: NIPSENSE - A Comparative Study of Nipple and Skin Sensation Preservation After Nipple-Sparing Mastectomy With Conventional, Endoscopic, and Robotic Techniques
Brief Title: A Comparative Study of Nipple Sensation Preservation After Nipple-Sparing Mastectomy With Conventional, Endoscopic, Robotic Techniques
Acronym: NIPSENSE
Status: Recruiting | Type: Observational
Sponsor: Candiolo Cancer Institute - IRCCS (Other)
Responsible Party: Principal Investigator, Giada Pozzi, MD, Candiolo Cancer Institute - IRCCS
Other Study IDs: NIPSENSE; 00043/2025 (Registry Identifier: Comitato Etico Città della Salute e della Scienza di Torino)
Record Dates: First submitted 2025-06-18; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Sensation Disorder
Keywords: Nipple sensation; Sensory outcomes; Quality of life; Endoscopic breast surgery; Robotic breast surgery; Breast cancer surgery; Nipple-sparing mastectomy; Breast reconstruction; R-NSM; E-NSM; conventional mastectomy
MeSH Terms: conditions — Sensation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conventional Nipple-Sparing Mastectomy (C-NSM): Participants in this group will undergo a standard open nipple-sparing mastectomy using traditional surgical instruments. The procedure is performed through a visible incision on the breast, while preserving the nipple and surrounding skin. An implant is placed for immediate reconstruction.
  Interventions: Diagnostic Test: Nipple Sensation Assessment
- Endoscopic Nipple-Sparing Mastectomy (E-NSM): This group will receive a minimally invasive nipple-sparing mastectomy using an endoscopic technique. The breast tissue is removed through a small incision in the armpit using a camera and specialized instruments. An implant is placed during the same surgery
  Interventions: Diagnostic Test: Nipple Sensation Assessment
- Robotic Nipple-Sparing Mastectomy (R-NSM): Participants in this group will undergo a robotic-assisted nipple-sparing mastectomy. The surgery is performed using a robotic surgical system through a small armpit incision, offering enhanced precision and visualization. Immediate implant reconstruction is also performed.
  Interventions: Diagnostic Test: Nipple Sensation Assessment

INTERVENTIONS:
Diagnostic Test: Nipple Sensation Assessment — the measurement of nipple sensation preservation, will be conducted using the Semmes-Weinstein esthesiometer. The clinician will use the device to touch the nipple and the surrounding quadrants of the skin, applying filaments of increasing calibers (0.07gr, 0.4gr, 2.0gr, 4.0gr, 300gr), and the lightest caliber perceived by the patient will be recorded. This assessment will be conducted at four different times:
  * Before surgery, to assess baseline sensation.
  * 1 month after surgery.
  * 3 months after surgery.
  * 6 months after surgery.

SUMMARY:
The goal of this comparative study is to learn how different surgical methods affect nipple and skin sensation after nipple-sparing mastectomy (NSM). The study will compare three types of NSM: conventional, endoscopic, and robotic.

The main question it aims to answer is:

How much nipple sensation do participants keep after each type of surgery?

Researchers will also look at surgery-related complications, patient-reported outcomes like body image and quality of life, and tissue analysis to see if there is a link between nerve structures and sensation.

Participants will:

Have NSM using one of the three surgical approaches

Receive breast reconstruction with an implant during the same surgery

Complete nipple sensation tests before and at 1, 3, and 6 months after surgery

Answer surveys about their quality of life and body image

Provide surgical tissue for analysis (as part of the planned procedure)

DETAILED DESCRIPTION:
The NIPSENSE study is a prospective, single-center study comparing how well nipple sensation is preserved after three types of nipple-sparing mastectomy (NSM): Conventional NSM (C-NSM), Endoscopic NSM (E-NSM), and Robotic NSM (R-NSM). The goal is to better understand the sensory and quality-of-life outcomes associated with each technique.

A total of 90 female participants (30 in each group) will be recruited. All will undergo NSM with direct-to-implant reconstruction. Participants will be assessed for nipple and skin sensation before surgery, and again at 1, 3, and 6 months after surgery, using a standard medical tool called the Semmes-Weinstein esthesiometer.

The study will also evaluate:

Surgical complications (e.g., infection, bleeding, skin necrosis)

Patient-reported outcomes using validated tools like the Hopwood Body Image Scale and EORTC questionnaires

Tissue analysis to explore whether preserved nerve structures are related to the level of sensation after surgery

This study will provide important data about how surgical methods impact physical and emotional outcomes for people undergoing mastectomy. The findings may help improve patient care and inform future decisions about surgical approaches to breast cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years.
* Diagnosed with early-stage breast cancer or deemed at high risk for breast cancer (eg. BRCA1-2 mutations).
* Candidates for Nipple-Sparing Mastectomy (NSM).
* Able to provide informed consent.
* No contraindications for surgery based on physical examination and preoperative assessment.
* Signed the consent forms and willing to participate in all scheduled follow-up assessments.

Exclusion Criteria:

* Previous breast surgery.
* History of radiation therapy to the chest/breast area.
* Active or non-controlled diabetes mellitus.
* Neuropathies causing potentially altered skin sensation.
* Nipple involvement by cancer, clinical or reported intra-operatively via frozen section analysis (the procedure will be converted to SSM).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of female patients aged 18 years or older, eligible for mastectomy for early-stage breast cancer or high-risk conditions, who meet the study eligibility criteria. A total of 90 patients will be recruited at Candiolo Cancer Institute in Torino (Italy).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
measurement of nipple sensation preservation | This assessment will be conducted at four different times: • Before surgery, to assess baseline sensation. • 1 month after surgery. • 3 months after surgery. • 6 months after surgery.
  The primary objective, the measurement of nipple sensation preservation, will be conducted using the Semmes-Weinstein esthesiometer. The clinician will use the device to touch the nipple and the surrounding quadrants of the skin, applying filaments of increasing calibers (0.07gr, 0.4gr, 2.0gr, 4.0gr, 300gr), and the lightest caliber perceived by the patient will be recorded.

SECONDARY OUTCOMES:
surgical outcomes | from enrollment to 3 months
  nipple-areola complex necrosis, skin flaps necrosis, infection, bleeding, seroma, wound dehiscence,
anatomopathological findings | 30-60 days post-surgery
  the presence or absence of sensory cutaneous receptors in the subcutaneous layer of the specimen and their possible correlation to the degree of cutaneous sensation
PROMs | From enrollment to 6 monts postoperatively
  Questionnaires will be administered to the patients to assess patient-reported outcomes: Hopwood Body Image Scale (score 0 to 30, higher scores meaning a worst outcome), and EORTC - European Organisation for Research and Treatment of Cancer, BR-23 questionnaire (no total score, each question compared individually between groups)

CONTACTS AND LOCATIONS:
Overall Officials: Giada Pozzi, MD, Principal Investigator — Candiolo Cancer Institute FPO-IRCCS
Locations (1):
- Candiolo Cancer Institute FPO-IRCCS, Torino, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available to qualified researchers upon reasonable request, following publication of the primary results. Shared data may include demographic details, surgical outcomes, complications, and patient-reported outcomes. Requests will be reviewed by the study team to ensure appropriate use and compliance with ethical standards. Data sharing will be subject to a data use agreement.
Supporting Information: CSR
Time Frame: IPD Sharing Time Frame: from 6 months to 24 months after end of recruitment
Access Criteria: Institutions involved in breast cancer research will be able to request access by directly contacting the PI and coordinating center of the study

REFERENCES:
- [Background] Moortgat P, Anthonissen M, Van Daele U, Meirte J, Vanhullebusch T, Maertens K. Objective Assessment Techniques: Physiological Parameters in Scar Assessment. 2020 Dec 8. In: Teot L, Mustoe TA, Middelkoop E, Gauglitz GG, editors. Textbook on Scar Management: State of the Art Management and Emerging Technologies [Internet]. Cham (CH): Springer; 2020. Chapter 18. Available from http://www.ncbi.nlm.nih.gov/books/NBK586121/ PMID 36351153
- [Background] Kostidou E, Schmelz M, Hasemaki N, Kokotis P. Objective Methods for Breast Sensibility Testing. Plast Reconstr Surg. 2019 Feb;143(2):398-404. doi: 10.1097/PRS.0000000000005200. PMID 30688881
- [Background] Tevlin R, Brazio P, Tran N, Nguyen D. Immediate targeted nipple-areolar complex re-innervation: Improving outcomes in immediate autologous breast reconstruction. J Plast Reconstr Aesthet Surg. 2021 Jul;74(7):1503-1507. doi: 10.1016/j.bjps.2020.11.021. Epub 2020 Dec 3. PMID 33341386
- [Background] Prado A, Andrades P, Benitez S, Parada F. Areola-nipple perception threshold to faradic electricity: a new measure of sensibility of the breasts. Aesthetic Plast Surg. 2008 Sep;32(5):748-52. doi: 10.1007/s00266-008-9148-4. Epub 2008 Apr 29. PMID 18443851
- [Background] Weinstein S. Fifty years of somatosensory research: from the Semmes-Weinstein monofilaments to the Weinstein Enhanced Sensory Test. J Hand Ther. 1993 Jan-Mar;6(1):11-22; discussion 50. PMID 8343870
- [Background] Santanelli F, Paolini G, Bittarelli D, Nofroni I. Computer-assisted evaluation of nipple-areola complex sensibility in macromastia and following superolateral pedicle reduction mammaplasty: a statistical analysis. Plast Reconstr Surg. 2007 May;119(6):1679-1683. doi: 10.1097/01.prs.0000258828.84107.59. PMID 17440341
- [Background] van Verschuer VM, Mureau MA, Gopie JP, Vos EL, Verhoef C, Menke-Pluijmers MB, Koppert LB. Patient Satisfaction and Nipple-Areola Sensitivity After Bilateral Prophylactic Mastectomy and Immediate Implant Breast Reconstruction in a High Breast Cancer Risk Population: Nipple-Sparing Mastectomy Versus Skin-Sparing Mastectomy. Ann Plast Surg. 2016 Aug;77(2):145-52. doi: 10.1097/SAP.0000000000000366. PMID 26076217
- [Background] Kasielska-Trojan A, Szulia A, Zawadzki T, Antoszewski B. The Assessment of Nipple Areola Complex Sensation with Semmes-Weinstein Monofilaments-Normative Values and Its Covariates. Diagnostics (Basel). 2021 Nov 19;11(11):2145. doi: 10.3390/diagnostics11112145. PMID 34829492
- [Background] Jerosch-Herold C. Assessment of sensibility after nerve injury and repair: a systematic review of evidence for validity, reliability and responsiveness of tests. J Hand Surg Br. 2005 Jun;30(3):252-64. doi: 10.1016/j.jhsb.2004.12.006. PMID 15862365
- [Background] Schlenz I, Kuzbari R, Gruber H, Holle J. The sensitivity of the nipple-areola complex: an anatomic study. Plast Reconstr Surg. 2000 Mar;105(3):905-9. doi: 10.1097/00006534-200003000-00012. PMID 10724249
- [Background] Bijkerk E, Cornelissen AJM, Sommer M, Van Der Hulst RRWJ, Lataster A, Tuinder SMH. Intercostal nerve block of the anterior cutaneous branches and the sensibility of the female breast. Clin Anat. 2020 Oct;33(7):1025-1032. doi: 10.1002/ca.23532. Epub 2019 Dec 23. PMID 31837172
- [Background] Riccio CA, Zeiderman MR, Chowdhry S, Brooks RM, Kelishadi SS, Tutela JP, Choo J, Yonick DV, Wilhelmi BJ. Plastic Surgery of the Breast: Keeping the Nipple Sensitive. Eplasty. 2015 Jul 2;15:e28. eCollection 2015. PMID 26171100
- [Background] Sarhadi NS, Shaw-Dunn J, Soutar DS. Nerve supply of the breast with special reference to the nipple and areola: Sir Astley Cooper revisited. Clin Anat. 1997;10(4):283-8. doi: 10.1002/(SICI)1098-2353(1997)10:43.0.CO;2-G. PMID 9213048
- [Background] Shridharani SM, Magarakis M, Stapleton SM, Basdag B, Seal SM, Rosson GD. Breast sensation after breast reconstruction: a systematic review. J Reconstr Microsurg. 2010 Jul;26(5):303-10. doi: 10.1055/s-0030-1249313. Epub 2010 Mar 1. PMID 20195965
- [Background] Rodriguez-Unda NA, Bello RJ, Clarke-Pearson EM, Sanyal A, Cooney CM, Manahan MA, Rosson GD. Nipple-Sparing Mastectomy Improves Long-Term Nipple But Not Skin Sensation After Breast Reconstruction: Quantification of Long-Term Sensation in Nipple Sparing Versus Non-nipple Sparing Mastectomy. Ann Plast Surg. 2017 Jun;78(6):697-703. doi: 10.1097/SAP.0000000000000900. PMID 27759590
- [Background] Peled AW, Amara D, Piper ML, Klassen AF, Tsangaris E, Pusic AL. Development and Validation of a Nipple-Specific Scale for the BREAST-Q to Assess Patient-Reported Outcomes following Nipple-Sparing Mastectomy. Plast Reconstr Surg. 2019 Apr;143(4):1010-1017. doi: 10.1097/PRS.0000000000005426. PMID 30921114
- [Background] Howard MA, Sisco M, Yao K, Winchester DJ, Barrera E, Warner J, Jaffe J, Hulick P, Kuchta K, Pusic AL, Sener SF. Patient satisfaction with nipple-sparing mastectomy: A prospective study of patient reported outcomes using the BREAST-Q. J Surg Oncol. 2016 Sep;114(4):416-22. doi: 10.1002/jso.24364. Epub 2016 Jul 8. PMID 27393183
- [Background] Benediktsson KP, Perbeck L, Geigant E, Solders G. Touch sensibility in the breast after subcutaneous mastectomy and immediate reconstruction with a prosthesis. Br J Plast Surg. 1997 Sep;50(6):443-9. doi: 10.1016/s0007-1226(97)90332-5. PMID 9326148
- [Background] Hammond JB, Kandi LA, Armstrong VL, Kosiorek HE, Rebecca AM, Casey WJ 3rd, Kruger EA, Cronin PA, Pockaj BA, Teven CM. Long-term breast and nipple sensation after nipple-sparing mastectomy with implant reconstruction: Relevance to physical, psychosocial, and sexual well-being. J Plast Reconstr Aesthet Surg. 2022 Sep;75(9):2914-2919. doi: 10.1016/j.bjps.2022.06.034. Epub 2022 Jun 20. PMID 35915018
- [Background] Dossett LA, Lowe J, Sun W, Lee MC, Smith PD, Jacobsen PB, Laronga C. Prospective evaluation of skin and nipple-areola sensation and patient satisfaction after nipple-sparing mastectomy. J Surg Oncol. 2016 Jul;114(1):11-6. doi: 10.1002/jso.24264. Epub 2016 Apr 18. PMID 27087574
- [Background] Shaffer K, Danko M, DeLaere A, Chant E, Pople B, Grisby S, Dekhne N. Patient satisfaction following nipple-sparing mastectomy and assessment of nipple-areolar sensation. Breast J. 2019 May;25(3):542-544. doi: 10.1111/tbj.13274. Epub 2019 Apr 18. No abstract available. PMID 31001911
- [Background] Gahm J, Hansson P, Brandberg Y, Wickman M. Breast sensibility after bilateral risk-reducing mastectomy and immediate breast reconstruction: a prospective study. J Plast Reconstr Aesthet Surg. 2013 Nov;66(11):1521-7. doi: 10.1016/j.bjps.2013.06.054. Epub 2013 Aug 13. PMID 23953096
- [Background] Akdeniz Dogan Z, Farhadi J. Evaluation of Sensation on Mastectomy Skin Flaps following Immediate Breast Reconstruction. J Reconstr Microsurg. 2020 Jul;36(6):420-425. doi: 10.1055/s-0040-1702157. Epub 2020 Feb 23. PMID 32088917
- [Background] Khan A, Zhang J, Sollazzo V, Mohammed K, Gui G. Sensory change of the reconstructed breast envelope after skin-sparing mastectomy. Eur J Surg Oncol. 2016 Jul;42(7):973-9. doi: 10.1016/j.ejso.2016.03.018. Epub 2016 Apr 9. PMID 27113424
- [Background] Laverdet B, Danigo A, Girard D, Magy L, Demiot C, Desmouliere A. Skin innervation: important roles during normal and pathological cutaneous repair. Histol Histopathol. 2015 Aug;30(8):875-92. doi: 10.14670/HH-11-610. Epub 2015 Mar 23. PMID 25799052
- [Background] Lai HW, Chang YL, Chandrachamnong K, See MH, Huang HI, Lin SL, Fang DY, Chen ST, Chen DR, Mok CW, Cheng FT. Factors associated with alteration of nipple or skin sensation and impact of duration of time following nipple-sparing mastectomy (NSM): an analysis of 460 cases with comparison of conventional versus endoscopic- or robotic-assisted NSM. World J Surg Oncol. 2023 Jul 26;21(1):222. doi: 10.1186/s12957-023-03107-5. PMID 37491239
- [Background] Bueno JN, Haddad CAS, Rizzi SKLA, Giron PS, Facina G, Nazario ACP. Evaluation of body image, quality of life, tactile sensitivity and pain in women with breast cancer submitted to surgical intervention. Rev Assoc Med Bras (1992). 2018 Jun;64(6):530-536. doi: 10.1590/1806-9282.64.06.530. PMID 30304311
- [Background] Barber R, Scheltens P, Gholkar A, Ballard C, McKeith I, Ince P, Perry R, O'Brien J. White matter lesions on magnetic resonance imaging in dementia with Lewy bodies, Alzheimer's disease, vascular dementia, and normal aging. J Neurol Neurosurg Psychiatry. 1999 Jul;67(1):66-72. doi: 10.1136/jnnp.67.1.66. PMID 10369824
- [Background] Lavery LA, Lavery DE, Lavery DC, Lafontaine J, Bharara M, Najafi B. Accuracy and durability of Semmes-Weinstein monofilaments: what is the useful service life? Diabetes Res Clin Pract. 2012 Sep;97(3):399-404. doi: 10.1016/j.diabres.2012.04.006. Epub 2012 May 3. PMID 22560793
- [Background] Longo B, Campanale A, Santanelli di Pompeo F. Nipple-areola complex cutaneous sensitivity: a systematic approach to classification and breast volume. J Plast Reconstr Aesthet Surg. 2014 Dec;67(12):1630-6. doi: 10.1016/j.bjps.2014.08.043. Epub 2014 Aug 27. PMID 25231086
- [Background] Bell-Krotoski J. Advances in sensibility evaluation. Hand Clin. 1991 Aug;7(3):527-46. PMID 1939358
- [Background] Jaspars JJ, Posma AN, van Immerseel AA, Gittenberger-de Groot AC. The cutaneous innervation of the female breast and nipple-areola complex: implications for surgery. Br J Plast Surg. 1997 Jun;50(4):249-59. doi: 10.1016/s0007-1226(97)91155-3. PMID 9215081
- [Background] Tairych GV, Kuzbari R, Rigel S, Todoroff BP, Schneider B, Deutinger M. Normal cutaneous sensibility of the breast. Plast Reconstr Surg. 1998 Sep;102(3):701-4. doi: 10.1097/00006534-199809030-00013. PMID 9727434
- See also: Institution Official Website — https://www.irccs.com/en